CLINICAL TRIAL: NCT06596343
Title: Study on the Value of Traditional Chinese Medicine Precision Treatment Based on Syndrome Differentiation in Postoperative Adjuvant Therapy for Locally Advanced Colorectal Cancer
Brief Title: Evaluating the Benefits of Personalized Traditional Chinese Medicine in Postoperative Treatment for Locally Advanced Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Zhangfa Song, Professor, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCM-1
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Locally Advanced Colorectal Cancer; Postoperative Adjuvant Therapy
MeSH Terms: interventions — Medicine, Chinese Traditional; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adjuvant Chemotherapy Combined with Traditional Chinese Medicine (TCM) Supportive Therapy (Experimental): Patients will sign an informed consent form after surgery but before starting chemotherapy, and those enrolled will receive a combination of chemotherapy and Traditional Chinese Medicine (TCM) supportive therapy.
  1. Chemotherapy Regimen:
     * Postoperative adjuvant chemotherapy: A dual-drug concurrent regimen will be used, with each cycle lasting 21 days. On day 1 of each cycle, oxaliplatin will be administered intravenously at a dose of 130 mg/m². From day 1 to day 14 of each cycle, capecitabine will be taken orally at a dose of 1000 mg/m², twice daily. The treatment duration will follow the CSCO 2023 guidelines for colorectal cancer, with chemotherapy lasting for 6 months.
  2. TCM Treatment:
     * TCM treatment will be based on syndrome differentiation ("Zheng") and guided by the Guidelines for TCM Diagnosis and Treatment of Malignant Tumors.
  Interventions: Drug: Adjuvant Chemotherapy Combined with Traditional Chinese Medicine (TCM) Supportive Therapy

INTERVENTIONS:
Drug: Adjuvant Chemotherapy Combined with Traditional Chinese Medicine (TCM) Supportive Therapy — 1. Chemotherapy Regimen:
     * Postoperative adjuvant chemotherapy: A dual-drug concurrent regimen will be used, with each cycle lasting 21 days. On day 1 of each cycle, oxaliplatin will be administered intravenously at a dose of 130 mg/m². From day 1 to day 14 of each cycle, capecitabine will be taken orally at a dose of 1000 mg/m², twice daily. The treatment duration will follow the CSCO 2023 guidelines for colorectal cancer, with chemotherapy lasting for 6 months.
  2. TCM Treatment:
     * TCM treatment will be based on syndrome differentiation ("Zheng") and guided by the Guidelines for TCM Diagnosis and Treatment of Malignant Tumors.

SUMMARY:
This study aims to explore the role of Traditional Chinese Medicine (TCM) based on syndrome differentiation in reducing chemotherapy side effects, lowering the risk of metastasis and recurrence, and improving survival rates in postoperative colorectal cancer patients through a prospective, single-arm interventional clinical trial.

DETAILED DESCRIPTION:
Colorectal cancer is the third leading cause of cancer-related deaths worldwide, with 1.9 million new cases and nearly 935,000 deaths reported in 2020. In China, colorectal cancer ranks third in new cases for both men and women, while it ranks fifth in cancer-related deaths among men and second among women. It has become a global public health issue and a major threat to people's health. Surgical resection is the primary treatment for colon cancer and can potentially cure the tumor. More than 50% of colon cancer patients are diagnosed at locally advanced stages (stage II and III). Even after curative surgery, about 50% of these patients experience tumor recurrence due to undetectable micrometastases that persist post-surgery. Most of these patients require adjuvant chemotherapy to eliminate micrometastases and improve cure rates. Postoperative adjuvant chemotherapy can eradicate hidden micrometastases and prolong survival in colorectal cancer patients. Large clinical trials have shown that adjuvant chemotherapy reduces the recurrence rate by 41% and overall mortality by 33%. Thus, surgery combined with postoperative adjuvant chemotherapy is the standard treatment approach to cure colon cancer.

However, about 25% of stage III colorectal cancer patients still relapse despite adjuvant chemotherapy, indicating that not all patients benefit from it. Additionally, postoperative adjuvant chemotherapy can cause numerous side effects. The IDEA study reported that grade 3 or higher chemotherapy-related toxicities occurred in 20% of patients receiving 3 months of adjuvant chemotherapy and 36.9% of patients receiving 6 months. These side effects include mucositis, vomiting, diarrhea, febrile neutropenia, fatigue, hair loss, hand-foot syndrome (pain, redness, and peeling of the skin on the palms and soles), neurotoxicity, and cardiotoxicity. The incidence and severity of these side effects vary depending on the specific drugs and administration methods, and some side effects, such as oxaliplatin-induced peripheral neuropathy, can persist long-term, significantly affecting patients' quality of life.

Thus, both healthcare providers and patients are seeking additional therapies to reduce toxicity and improve the efficacy of standard treatment. In real-world practice, many colorectal cancer patients have received Traditional Chinese Medicine (TCM) as part of their postoperative care, and TCM plays a significant role in colorectal cancer prevention and treatment.

In TCM, colorectal cancer is classified under conditions such as "zang du" (organ toxin), "chang ji" (intestinal accumulation), and "ji ju" (mass accumulation), primarily caused by irregular diet, emotional imbalance, and deficiency of vital energy (qi). Although the disease originates in the intestines, it is closely related to the spleen, stomach, liver, and kidneys. Early-stage disease is dominated by damp-heat and toxin stagnation, while later stages are characterized by a deficiency of vital energy with excess pathogenic factors, typically involving spleen and kidney yang deficiency, qi and blood deficiency, or liver and kidney yin deficiency. A deficiency in vital energy and yin-yang imbalance are key factors in the development of colorectal cancer. Damp-heat accumulation in the intestines leads to stagnation of qi, toxin formation, and eventual mass formation, which is a core mechanism of disease development.

This study aims to investigate the role of adding TCM during and after surgery and chemotherapy to enhance the clinical efficacy of adjuvant chemotherapy, reduce the occurrence of adverse effects, prevent metastasis and recurrence, and ultimately improve survival rates.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 18 and 75 years. 2. Diagnosed with colorectal cancer at Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, and underwent standard radical colorectal cancer surgery. Postoperative pathological staging is stage III (AJCC 8th edition: T4, any N+, M0, or any T, N2, M0), indicating the need for chemotherapy according to the CSCO 2023 colorectal cancer guidelines.

  3. Willing to receive Traditional Chinese Medicine (TCM) treatment. 4. Voluntarily agree to participate in the study and sign the informed consent form. If the subject is unable to read or sign the consent due to incapacity, the informed consent must be obtained from a legal guardian. If the subject cannot read the consent (e.g., illiterate subjects), a witness must observe and sign the consent process.

  5. Expected survival of ≥12 months. 6. ECOG performance status score of 0-1. 7. No prior anti-cancer, immunotherapy, or radiation treatment. 8. Laboratory tests meeting the following criteria:
* White blood cell count ≥3.5 × 10^9/L, absolute neutrophil count ≥1.8 × 10^9/L, platelet count ≥100 × 10^9/L, hemoglobin ≥100 g/L.
* INR ≤1.5 and APTT ≤1.5 times the upper limit of normal (ULN) or PTT ≤1.5 times ULN.
* Total bilirubin ≤1.25 times ULN; ALT and AST ≤3 times ULN; serum albumin ≥28 g/L.
* 24-hour creatinine clearance rate ≥50 mL/min or serum creatinine ≤1.5 times ULN.

Exclusion Criteria:

* 1. Colorectal cancer patients with distant metastasis as indicated by preoperative evaluation.

  2. Postoperative pathological results indicate that chemotherapy is not required according to the CSCO 2023 colorectal cancer guidelines.

  3. Patients who have received neoadjuvant chemoradiotherapy before surgery. 4. Patients with severe heart, liver, kidney damage, or bone marrow dysfunction.

  5. Pregnant or breastfeeding women. 6. Patients with known allergies to Traditional Chinese Medicine components. 7. Patients who refuse chemotherapy or TCM treatment. 8. Patients with a history of mental illness or cognitive impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade III/IV adverse events | From the beginning of the first chemotherapy to three months after the end of the course of chemotherapy
  According to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, adverse events (AEs) are graded on a scale from 1 to 5 based on severity:
  * Grade I: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; no intervention required.
  * Grade II: Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADLs).
  * Grade III: Severe; medically significant but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated; disabling; limiting self-care ADLs.
  * Grade IV: Life-threatening consequences; urgent intervention required.
  * Grade V: Death related to adverse event.

SECONDARY OUTCOMES:
3-year Disease-Free Survival | 3 years post-treatment
  3-year Disease-Free Survival (DFS) refers to the percentage of patients who remain free from any signs or symptoms of cancer recurrence or progression for three years after treatment.
3-year Overall Survival | 3 years post-treatment
  3-year Overall Survival (OS) refers to the percentage of patients who are still alive three years after the start of treatment, regardless of whether the cancer has recurred or progressed.
Completion rate of adjuvant chemotherapy | From the beginning of the first chemotherapy to the end of the course of chemotherapy, up to 6 months.
  The completion rate of adjuvant chemotherapy is defined as the percentage of patients who successfully complete the full chemotherapy regimen within 6 months post-surgery, in accordance with the CSCO 2023 guidelines for colorectal cancer
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 | From the beginning of the first chemotherapy to three months after the end of the course of chemotherapy
  The EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) is a widely used tool for assessing the quality of life of cancer patients in clinical trials. Each subscale of the EORTC QLQ-C30 is scored on a range from 0 to 100. Score Interpretation: Higher Scores:
  For functional scales (e.g., physical, role, emotional, cognitive, social functioning): Higher scores indicate a better quality of life. For symptom scales (e.g., fatigue, pain, nausea/vomiting): Higher scores indicate worse symptoms or problems.
  The global health status/QoL scale: Higher scores indicate a better overall quality of life.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Colorectal Cancer Module （EORTC QLQ-CR29） | From the beginning of the first chemotherapy to three months after the end of the course of chemotherapy
  The EORTC QLQ-CR29 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Colorectal Cancer Module) is a supplementary tool to the EORTC QLQ-C30, specifically designed to assess the quality of life in patients with colorectal cancer. Similar to the EORTC QLQ-C30, each item or subscale in the EORTC QLQ-CR29 is scored on a scale of 0 to 100.
  Score Interpretation: Higher Scores: For functional scales (e.g., body image, sexual functioning): Higher scores reflect better functioning and, thus, a better quality of life. For symptom scales (e.g., bowel symptoms, urinary symptoms, blood/mucus in stool): Higher scores indicate worse symptoms, reflecting a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou, China, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grothey A, Sobrero AF, Shields AF, Yoshino T, Paul J, Taieb J, Souglakos J, Shi Q, Kerr R, Labianca R, Meyerhardt JA, Vernerey D, Yamanaka T, Boukovinas I, Meyers JP, Renfro LA, Niedzwiecki D, Watanabe T, Torri V, Saunders M, Sargent DJ, Andre T, Iveson T. Duration of Adjuvant Chemotherapy for Stage III Colon Cancer. N Engl J Med. 2018 Mar 29;378(13):1177-1188. doi: 10.1056/NEJMoa1713709. PMID 29590544
- [Background] Taghizadeh H, Prager GW. Personalized Adjuvant Treatment of Colon Cancer. Visc Med. 2020 Oct;36(5):397-406. doi: 10.1159/000508175. Epub 2020 Jun 29. PMID 33178737
- [Background] Sauer S, Reed DR, Ihnat M, Hurst RE, Warshawsky D, Barkan D. Innovative Approaches in the Battle Against Cancer Recurrence: Novel Strategies to Combat Dormant Disseminated Tumor Cells. Front Oncol. 2021 Apr 27;11:659963. doi: 10.3389/fonc.2021.659963. eCollection 2021. PMID 33987095
- [Background] Nelson H, Petrelli N, Carlin A, Couture J, Fleshman J, Guillem J, Miedema B, Ota D, Sargent D; National Cancer Institute Expert Panel. Guidelines 2000 for colon and rectal cancer surgery. J Natl Cancer Inst. 2001 Apr 18;93(8):583-96. doi: 10.1093/jnci/93.8.583. PMID 11309435
- [Background] Siegel RL, Wagle NS, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2023. CA Cancer J Clin. 2023 May-Jun;73(3):233-254. doi: 10.3322/caac.21772. Epub 2023 Mar 1. PMID 36856579